CLINICAL TRIAL: NCT07309536
Title: Mediterranean Diet Uptake and Nutrition on Child Health, Inflammation, and Early-life Symbiosis (MUNCHIES): A Randomized Controlled Trial
Brief Title: Mediterranean Diet Uptake and Nutrition on Child Health, Inflammation, and Early-life Symbiosis (MUNCHIES) Study
Acronym: MUNCHIES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Brunswick (Other)
Responsible Party: Principal Investigator, Maryam Kebbe, Associate Professor, University of New Brunswick
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB 2025-146
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Gut Microbiome; Body Composition; Adherence; Metabolites; Inflammation
Keywords: Dietary patterns; Gastrointestinal microbiome; Body composition; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet Intervention (Experimental): Toddlers in this group will follow a Mediterranean-style diet for nine weeks. Families will receive Mediterranean diet foods for three weeks and take part in nine weekly sessions (one overview and eight follow-up sessions) focused on preparing toddler-appropriate Mediterranean meals. The sessions are designed to support consistency in feeding, track progress, and provide guidance on diet adherence. Measurements of toddler height, weight, body composition (BOD POD), stool samples, and questionnaires will be collected at baseline, 3 weeks, and 3 months post-baseline.
  Interventions: Behavioral: Mediterranean Diet Nutrition Program
- Standard Diet (Active Comparator): Toddlers in this group will continue their usual diets for nine weeks while families participate in nine weekly general nutrition education sessions. Measurements of toddler height, weight, body composition (BODPOD), stool samples, and questionnaires will occur at the same time points as the intervention group. Families in this group will receive a $100 honorarium.
  Interventions: Behavioral: Standard Diet Education Program

INTERVENTIONS:
Behavioral: Mediterranean Diet Nutrition Program — A nine session nutrition and feeding program designed to assess how a Mediterranean-style diet influences toddler gut health, body composition, and inflammation. Toddlers will receive Mediterranean-style foods for the first three weeks, followed by continued guidance through bi-weekly educational sessions focused on meal preparation, food variety, and adherence. Specifically sessions will cover key topics such as toddler nutrient needs, budget-friendly meal planning, picky eating, family mealtime strategies, and mindful eating. The program emphasizes incorporating fruits, vegetables, legumes, whole grains, and healthy fats into toddler meals, reducing ultra-processed foods, and promoting balanced feeding during early childhood.
  Arms: Mediterranean Diet Intervention
Behavioral: Standard Diet Education Program — A nine session general toddler nutrition education program designed to reflect typical dietary patterns in Canadian families. Families receive sessions on topics such as feeding styles, cultural foods and feeding practices, understanding nutrition labels, food safety, choking hazards and prevention, healthy recipes, myths and misinformation, and meal structure and routines. No study foods are provided. Toddlers maintain their usual diets throughout the study while completing the same measurements as those in the intervention group.
  Arms: Standard Diet

SUMMARY:
Toddlerhood (ages 2-3) is a critical window when the gut microbiome is still developing and eating habits are being established. Yet, many Canadian toddlers eat diets high in sugar and salt, which may affect long-term health. This study will test whether a MED diet can improve dietary inflammation, gut health, and body composition in toddlers and whether a tailored nutrition education program for parents can help families maintain healthy eating patterns.

In this study, toddlers will be randomly assigned to a 3-week MED diet or their usual diet. Families in the MED diet group will receive free meal boxes for the 3 weeks, plus guidance from a nutrition researcher through a structured education program. The standard diet group will continue their regular diet with general nutrition advice. Researchers will collect dietary information, body composition assessments, and stool samples to measure gut microbiome composition and metabolites.

This first study of a controlled diet intervention in toddlers, combining behavioral support, high-quality food provision, and advanced gut microbiome analysis, will help understand how early diet shapes lifelong eating habits and health, guiding public health strategies and precision nutrition approaches to prevent chronic disease from early life.

DETAILED DESCRIPTION:
The gut microbiome, central to immune and metabolic regulation, is highly responsive to dietary inputs. In adults, interventions like the Mediterranean (MED) diet rapidly increase beneficial microbial taxa and anti-inflammatory metabolites. Toddlerhood (24-36 months) represents a critical window when the gut microbiome continues to stabilize and dietary patterns become established. Yet, the diets of Canadian toddlers remain suboptimal, often dominated by high-sodium, high-sugar foods.

The aims of this study are to determine the effects of a (i) MED diet food-provision intervention on dietary inflammation, the gut microbiome and metabolites, and body composition of toddlers aged 2-3 years at 3 weeks and (ii) comprehensive, tailored nutrition education program, with or without food provision, in promoting adherence to the prescribed diets at 3 weeks and 3 months post-baseline.

This parallel randomized controlled trial at the University of New Brunswick will randomized parent-toddler dyads to either a 3-week MED diet or a Standard diet. Families in the MED diet group will receive free food provision and a tailored, theory-driven parental nutrition program. They will be provided with packaged food boxes including three meals (breakfast/lunch/dinner) and two snacks for each day of the week. Meals will be developed and prepared by a registered dietitian in UNB's metabolic kitchen under sterile conditions and delivered to parents in coolers. Families in the Standard diet group will continue to consume their regular diet and receive general nutrition education. Both groups will be initially screened using the KIDMED 2.0 to ensure they do not already adopt a MED diet. The nutrition education programs will be delivered over a 3-month period from baseline.

The primary outcome is the between-group difference in Children's Dietary Inflammatory Index scores at 3 weeks, diet adherence, and program satisfaction. Secondary outcomes include microbial diversity, taxa, metabolite profiles, body composition, blood pressure, and additional feeding metrics. Assessments will occur at baseline, 3 weeks, and 3 months. Stool samples will be analyzed using shallow shotgun metagenomics and metabolomics to assess microbial taxa, SCFAs, and other metabolites. Statistical analyses, conducted in R, will include t-tests, PERMANOVA, and mediation models.

The toddler years are a pivotal time for shaping lifelong eating habits and health outcomes, persisting into adolescence and adulthood. This is the first trial to test a controlled dietary intervention in toddlers, integrating behavioural theory and patient-oriented research. It will bring together a multifaceted team, combining expertise in nutrition and dietetics with cutting-edge knowledge in genomics for gut microbiome analysis. Findings will inform public health strategies and advance precision nutrition to reduce chronic disease risk from early life.

ELIGIBILITY:
Inclusion Criteria:

* Parent is ≥19 years of age.
* Carried a singleton pregnancy.
* Delivered at term (≥37 weeks gestation).
* Delivered vaginally or by cesarean section.
* Infant was born with a birth weight between 2,500 g and 4,500 g.
* Toddler is between 24 and 36 months of age at enrollment.
* Parent is able to communicate in English.
* Parent is willing to adhere to the Mediterranean diet for their toddler for 3 weeks.
* Parent is willing to participate in a nutrition education program for 3 months.
* Parent is willing to complete all measurements and provide a stool sample from their toddler.

Exclusion Criteria:

* Toddler has food allergies or dietary restrictions (e.g., gluten-free) that make it difficult to follow a Mediterranean diet.
* Toddler is at high risk for food allergies (e.g., strong family history of multiple food allergies common to the Mediterranean diet).
* Toddler is already following a Mediterranean diet.
* Toddler has had recent or active consumption of antibiotics, probiotics, or prebiotic drops.
* Toddler has an active acute illness, such as fever, diarrhea, or constipation.
* Toddler was born with a congenital illness or malformation that could affect diet, inflammation, gut health, or body composition.
* Toddler is currently breastfeeding, formula-feeding, or combination feeding.

Ages: 24 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Mediterranean Diet Adherence | Baseline, at 3 weeks, and at 3 months after enrollment.
  Adherence to the Mediterranean diet will be defined as the degree to which toddlers' and parents' food intake aligns with core Mediterranean diet principles (high intake of fruits, vegetables, legumes, whole grains, fish, and healthy fats; limited red meat, processed foods, and added sugars). Adherence will be assessed using the KIDMED 2.0 questionnaire for toddlers and a validated Mediterranean Diet Adherence Screener (MEDAS) for parents, weekly for the first 3 weeks and every two weeks for the remaining 9 weeks. Scores range from 0 to 12 for toddlers and 0 to 14 for parents, with higher scores indicating greater adherence.
Program Feasibility and Acceptability | Ongoing throughout study (baseline to 3 months).
  Feasibility will be assessed via recruitment, retention, adherence to diet, attendance at nutrition sessions, and completion of study measures. Acceptability will be assessed through parent-reported satisfaction surveys regarding the diet and education program.
Children's Dietary Inflammatory Index (C-DII) | Baseline, at 3 weeks, and at 3 months after enrollment.
  The Children's Dietary Inflammatory Index (C-DII) quantifies the inflammatory potential of an individual's diet. For this study, toddler dietary intake obtained from 24-hour dietary recalls (one weekday and one weekend per week for first 3 weeks, every two weeks for final 9 weeks) will be used to calculate C-DII scores. The DII scoring algorithm assigns weights to nutrient and food component intake based on their established inflammatory properties. Higher DII scores indicate more pro-inflammatory dietary patterns, whereas lower (more negative) scores represent more anti-inflammatory diets aligned with Mediterranean-style eating.

SECONDARY OUTCOMES:
Gut Microbiome Diversity, Composition, and Metabolites | Baseline, at 3 weeks, and at 3 months after enrollment.
  Gut microbiome diversity and taxa will be assessed using metagenomic sequencing of stool samples collected from toddlers. Alpha diversity metrics (e.g., Shannon index, Chao1) and beta diversity metrics (Bray-Curtis dissimilarity) will quantify within- and between-sample microbial diversity. Taxonomic composition at phylum, family, and genus levels will also be examined, as well as microbial metabolite profiles relevant to inflammation and metabolic regulation.
Toddler Anthropometrics, Body Composition, and Blood Pressure | Baseline, at 3 weeks, and at 3 months after enrollment.
  Toddler growth and body composition will be assessed using standardized anthropometric and air-displacement plethysmography methods. Height and weight will be measured to calculate body mass index (BMI), which will then be converted to BMI-for-age percentiles and/or z-scores using WHO growth standards to characterize growth status. Waist circumference will be collected. Body composition will be evaluated using the BOD POD Pediatric Option, an air-displacement plethysmography system that provides estimates of fat mass, fat-free mass, and percentages. Together, these metrics will provide data on dietary patterns may impact growth and body composition. Blood pressure will be measured using a manual sphygmomanometer, which will provide additional indication of cardiovascular health and risk for hypertension-related conditions.
Nutrition-Related Behaviors and Feeding Practices | Baseline, at 3 weeks, and at 3 months after enrollment.
  Parents' feeding practices and toddlers' eating behaviors will be assessed using validated self-report questionnaires, such as the Child Feeding Questionnaire (CFQ) and the Feeding Practices and Structure Questionnaire (FPSQ). Each instrument generates subscale scores by averaging item responses within each domain. For the CFQ, items are rated on 1-5 Likert scales, and subscales such as Restriction, Pressure to Eat, and Monitoring are calculated by averaging item scores; higher values indicate greater use of that feeding practice. For the FPSQ, items are also scored on Likert scales and grouped into Structure (e.g., routines, limits) and Autonomy Support (e.g., encouragement, involvement) subscales, with mean scores reflecting how frequently each practice is used. These procedures quantify parental control, responsiveness, feeding structure, and child eating behaviors (e.g., neophobia, appetite traits), offering a multidimensional profile of feeding dynamics.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Maryam Kebbe, PhD, CLC, Principal Investigator — University of New Brunswick
Locations (1):
- University of New Brunswick, Fredericton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kheirmandparizi M, Gouin JP, Bouchaud CC, Kebbe M, Bergeron C, Madani Civi R, Rhodes RE, Farnesi BC, Bouguila N, Conklin AI, Lear SA, Cohen TR. Perceptions of self-monitoring dietary intake according to a plate-based approach: A qualitative study. PLoS One. 2023 Nov 28;18(11):e0294652. doi: 10.1371/journal.pone.0294652. eCollection 2023. PMID 38015899
- [Background] Kebbe M, Leung K, Perrett B, Reimer RA, Adamo K, Redman LM. Effects of Infant Formula Supplemented With Prebiotics on the Gut Microbiome, Gut Environment, Growth Parameters, and Safety and Tolerance: A Systematic Review and Meta-Analysis. Nutr Rev. 2025 Mar 1;83(3):422-447. doi: 10.1093/nutrit/nuae184. PMID 39832301
- [Background] Redman LM, Phelan S, Apolzan JW, Beyl RA, Altazan AD, Dickey MS, Simeon E, Flanagan EW, Cabre HE, Sparks JR, Kebbe M, Caughey AB, Valent AM, Hsia DS, Yin E, Keadle SK. Protocol for a randomised controlled trial of a weight maintenance intervention to promote fat loss in pregnant individuals with obesity. BMJ Open. 2025 Feb 25;15(2):e095804. doi: 10.1136/bmjopen-2024-095804. PMID 40000086
- [Background] Kebbe M, Eaton A, Dyson M, Scott S, McHUGH T, Yaskina M, Ladha T, Islam B, Talwar K, Wincott J, Ball G. Testing the Feasibility, User Experiences, and Preliminary Effect of Conversation Cards for Adolescents(c) For Behavior Change and Collaborative Goal Setting in Primary Care: A Pilot Randomized Controlled Trial. J Health Commun. 2024 Oct 2;29(10):663-671. doi: 10.1080/10810730.2024.2411318. Epub 2024 Oct 7. PMID 39374045
- [Background] Song X, Yang K, Cheng C, Hu Q, Zhao F, Lu S, Long J, Yang H, Chen S. Higher dietary inflammatory index linked to increased risk of hypertension: a systematic review and dose-response meta-analysis. Eur J Clin Nutr. 2025 Jun;79(6):512-519. doi: 10.1038/s41430-024-01530-9. Epub 2024 Oct 24. PMID 39448814
- [Background] Chen GQ, Peng CL, Lian Y, Wang BW, Chen PY, Wang GP. Association Between Dietary Inflammatory Index and Mental Health: A Systematic Review and Dose-Response Meta-Analysis. Front Nutr. 2021 May 5;8:662357. doi: 10.3389/fnut.2021.662357. eCollection 2021. PMID 34026809
- [Background] Liu FH, Liu C, Gong TT, Gao S, Sun H, Jiang YT, Zhang JY, Zhang M, Gao C, Li XY, Zhao YH, Wu QJ. Dietary Inflammatory Index and Health Outcomes: An Umbrella Review of Systematic Review and Meta-Analyses of Observational Studies. Front Nutr. 2021 May 19;8:647122. doi: 10.3389/fnut.2021.647122. eCollection 2021. PMID 34095187
- [Background] Mayr HL, Thomas CJ, Tierney AC, Kucianski T, George ES, Ruiz-Canela M, Hebert JR, Shivappa N, Itsiopoulos C. Randomization to 6-month Mediterranean diet compared with a low-fat diet leads to improvement in Dietary Inflammatory Index scores in patients with coronary heart disease: the AUSMED Heart Trial. Nutr Res. 2018 Jul;55:94-107. doi: 10.1016/j.nutres.2018.04.006. Epub 2018 Apr 14. PMID 29754829
- [Background] Hurley KM, Pepper MR, Candelaria M, Wang Y, Caulfield LE, Latta L, Hager ER, Black MM. Systematic development and validation of a theory-based questionnaire to assess toddler feeding. J Nutr. 2013 Dec;143(12):2044-9. doi: 10.3945/jn.113.179846. Epub 2013 Sep 25. PMID 24068792
- [Background] Moroney C, O'Leary F, Flood VM. The Med-NKQ: A Reliable Mediterranean Diet Nutrition Knowledge Questionnaire for Cardiovascular Disease. Nutrients. 2021 Aug 25;13(9):2949. doi: 10.3390/nu13092949. PMID 34578825
- [Background] Zongrone AA, Menon P, Pelto GH, Habicht JP, Rasmussen KM, Constas MA, Vermeylen F, Khaled A, Saha KK, Stoltzfus RJ. The Pathways from a Behavior Change Communication Intervention to Infant and Young Child Feeding in Bangladesh Are Mediated and Potentiated by Maternal Self-Efficacy. J Nutr. 2018 Feb 1;148(2):259-266. doi: 10.1093/jn/nxx048. PMID 29490102
- [Background] Wang Z, Bergeron N, Levison BS, Li XS, Chiu S, Jia X, Koeth RA, Li L, Wu Y, Tang WHW, Krauss RM, Hazen SL. Impact of chronic dietary red meat, white meat, or non-meat protein on trimethylamine N-oxide metabolism and renal excretion in healthy men and women. Eur Heart J. 2019 Feb 14;40(7):583-594. doi: 10.1093/eurheartj/ehy799. PMID 30535398
- [Background] Beckman JA, Shibao CA. Trimethylamine-N-Oxide, More Red Meat for the Vascular Scientists. Hypertension. 2020 Jul;76(1):40-41. doi: 10.1161/HYPERTENSIONAHA.120.14857. Epub 2020 Jun 10. No abstract available. PMID 32520618
- [Background] Leung AK, Marchand V, Sauve RS; Canadian Paediatric Society, Nutrition and Gastroenterology Committee. The 'picky eater': The toddler or preschooler who does not eat. Paediatr Child Health. 2012 Oct;17(8):455-60. doi: 10.1093/pch/17.8.455. PMID 24082809
- [Background] Davis C, Bryan J, Hodgson J, Murphy K. Definition of the Mediterranean Diet; a Literature Review. Nutrients. 2015 Nov 5;7(11):9139-53. doi: 10.3390/nu7115459. PMID 26556369
- [Background] Homann CM, Rossel CAJ, Dizzell S, Bervoets L, Simioni J, Li J, Gunn E, Surette MG, de Souza RJ, Mommers M, Hutton EK, Morrison KM, Penders J, van Best N, Stearns JC. Infants' First Solid Foods: Impact on Gut Microbiota Development in Two Intercontinental Cohorts. Nutrients. 2021 Jul 30;13(8):2639. doi: 10.3390/nu13082639. PMID 34444798
- [Background] Lopez-Gajardo MA, Leo FM, Sanchez-Miguel PA, Lopez-Gajardo D, Soulas C, Tapia-Serrano MA. KIDMED 2.0, An update of the KIDMED questionnaire: Evaluation of the psychometric properties in youth. Front Nutr. 2022 Nov 8;9:945721. doi: 10.3389/fnut.2022.945721. eCollection 2022. PMID 36424923
- [Background] Khan S, Wirth MD, Ortaglia A, Alvarado CR, Shivappa N, Hurley TG, Hebert JR. Design, Development and Construct Validation of the Children's Dietary Inflammatory Index. Nutrients. 2018 Jul 30;10(8):993. doi: 10.3390/nu10080993. PMID 30061487
- [Background] Downs SM, Willows ND. Should Canadians eat according to the traditional Mediterranean diet pyramid or Canada's food guide? Appl Physiol Nutr Metab. 2008 Jun;33(3):527-35. doi: 10.1139/H08-030. PMID 18461106
- [Background] de Franchis R, Bozza L, Canale P, Chiacchio M, Cortese P, D'Avino A, De Giovanni M, Iacovo MD, D'Onofrio A, Federico A, Gasparini N, Iaccarino F, Romano G, Spadaro R, Tedesco M, Vitiello G, Antignani A, Auricchio S, Valentino V, De Filippis F, Ercolini D, Bruzzese D. The Effect of Weaning with Adult Food Typical of the Mediterranean Diet on Taste Development and Eating Habits of Children: A Randomized Trial. Nutrients. 2022 Jun 15;14(12):2486. doi: 10.3390/nu14122486. PMID 35745216
- [Background] Hack S, Jessri M, L'Abbe MR. Nutritional quality of the food choices of Canadian children. BMC Nutr. 2021 May 29;7(1):16. doi: 10.1186/s40795-021-00422-6. PMID 34049592
- [Background] Birch L, Savage JS, Ventura A. Influences on the Development of Children's Eating Behaviours: From Infancy to Adolescence. Can J Diet Pract Res. 2007;68(1):s1-s56. No abstract available. PMID 19430591
- [Background] Fernandez-Jimenez R, Al-Kazaz M, Jaslow R, Carvajal I, Fuster V. Children Present a Window of Opportunity for Promoting Health: JACC Review Topic of the Week. J Am Coll Cardiol. 2018 Dec 25;72(25):3310-3319. doi: 10.1016/j.jacc.2018.10.031. Epub 2018 Dec 6. PMID 30527619
- [Background] Sarkar A, Yoo JY, Valeria Ozorio Dutra S, Morgan KH, Groer M. The Association between Early-Life Gut Microbiota and Long-Term Health and Diseases. J Clin Med. 2021 Jan 25;10(3):459. doi: 10.3390/jcm10030459. PMID 33504109
- [Background] Wernroth ML, Peura S, Hedman AM, Hetty S, Vicenzi S, Kennedy B, Fall K, Svennblad B, Andolf E, Pershagen G, Theorell-Haglow J, Nguyen D, Sayols-Baixeras S, Dekkers KF, Bertilsson S, Almqvist C, Dicksved J, Fall T. Development of gut microbiota during the first 2 years of life. Sci Rep. 2022 May 31;12(1):9080. doi: 10.1038/s41598-022-13009-3. PMID 35641542
- [Background] Bourdeau-Julien I, Castonguay-Paradis S, Rochefort G, Perron J, Lamarche B, Flamand N, Di Marzo V, Veilleux A, Raymond F. The diet rapidly and differentially affects the gut microbiota and host lipid mediators in a healthy population. Microbiome. 2023 Feb 11;11(1):26. doi: 10.1186/s40168-023-01469-2. PMID 36774515
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Background] Tilg H, Moschen AR. Food, immunity, and the microbiome. Gastroenterology. 2015 May;148(6):1107-19. doi: 10.1053/j.gastro.2014.12.036. Epub 2015 Jan 6. PMID 25575570
- [Background] Bujtor M, Turner AI, Torres SJ, Esteban-Gonzalo L, Pariante CM, Borsini A. Associations of Dietary Intake on Biological Markers of Inflammation in Children and Adolescents: A Systematic Review. Nutrients. 2021 Jan 25;13(2):356. doi: 10.3390/nu13020356. PMID 33503979
- [Background] Furman D, Campisi J, Verdin E, Carrera-Bastos P, Targ S, Franceschi C, Ferrucci L, Gilroy DW, Fasano A, Miller GW, Miller AH, Mantovani A, Weyand CM, Barzilai N, Goronzy JJ, Rando TA, Effros RB, Lucia A, Kleinstreuer N, Slavich GM. Chronic inflammation in the etiology of disease across the life span. Nat Med. 2019 Dec;25(12):1822-1832. doi: 10.1038/s41591-019-0675-0. Epub 2019 Dec 5. PMID 31806905
- [Background] Bach AM, Xie W, Piazzoli L, Jensen SKG, Afreen S, Haque R, Petri WA, Nelson CA. Systemic inflammation during the first year of life is associated with brain functional connectivity and future cognitive outcomes. Dev Cogn Neurosci. 2022 Feb;53:101041. doi: 10.1016/j.dcn.2021.101041. Epub 2021 Dec 7. PMID 34973509
- [Background] Sen S, Rifas-Shiman SL, Shivappa N, Wirth MD, Hebert JR, Gold DR, Gillman MW, Oken E. Associations of prenatal and early life dietary inflammatory potential with childhood adiposity and cardiometabolic risk in Project Viva. Pediatr Obes. 2018 May;13(5):292-300. doi: 10.1111/ijpo.12221. Epub 2017 May 10. PMID 28493362
- [Background] Palmer ER, Morales-Munoz I, Perry BI, Marwaha S, Warwick E, Rogers JC, Upthegrove R. Trajectories of Inflammation in Youth and Risk of Mental and Cardiometabolic Disorders in Adulthood. JAMA Psychiatry. 2024 Nov 1;81(11):1130-1137. doi: 10.1001/jamapsychiatry.2024.2193. PMID 39167392
- See also: Kebbe M. Nutribiomes Youtube Channel. — https://www.youtube.com/@nutribiomes
- See also: CMAJ. Patient-Oriented Research Collection. — https://www.cmajopen.ca/patient-oriented-research
- See also: World Health Organization. (2018). Noncommunicable diseases fact sheet. — https://www.who.int/news-room/fact-sheets/detail/noncommunicable-diseases
- See also: Statistics Canada. (2020). Leading causes of death, total population, by age group. Accessed August 20, 2024. — https://www150.statcan.gc.ca/t1/tbl1/en/tv.action?pid=1310039401